CLINICAL TRIAL: NCT04337437
Title: The Phase I Clinical Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Genakumab for Injection in Chinese Healthy Volunteers
Brief Title: Clinical Study of Genakumab for Injection in Chinese Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GenSci 048-I CT
Record Dates: First submitted 2020-04-01; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind (participant, investigator), excluding one non-blind investigator doctor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genakumab injection：5 groups (Experimental): 150 mg/1ml/bottle, single subcutaneous injection. Group A : 0.3mg/kg, Group B : 1mg/kg, Group C : 2mg/kg, Group D：4mg/kg, Group E : 6mg/kg,
  Interventions: Drug: Genakumab
- Placebo for this trial : 5 groups (Placebo Comparator): The placebo contains other excipients except Genakumab, and its appearance is consistent with that of Genakumab for injection, 150 mg/1ml/bottle, single subcutaneous injection.
  Group A : 0.3mg/kg, Group B : 1mg/kg, Group C : 2mg/kg, Group D：4mg/kg, Group E : 6mg/kg,
  Interventions: Drug: Placebo for this trial

INTERVENTIONS:
Drug: Genakumab — 150 mg/1ml/bottle, single subcutaneous injection.
  Arms: Genakumab injection：5 groups
Drug: Placebo for this trial — The placebo contains other excipients except Genakumab, and its appearance is consistent with that of Genakumab for injection, 150 mg/1ml/bottle, single subcutaneous injection.
  Arms: Placebo for this trial : 5 groups

SUMMARY:
To evaluate the safety and tolerability of single subcutaneous injection of Genakumab for Injection in Chinese healthy adult volunteers

DETAILED DESCRIPTION:
There are 5 dose groups with 8 participants in each group, including 6 participants in the experimental group and 2 participants in the placebo control group.

Since the strength of experimental drug is 150mg/1ml/ bottle, participants with a single dose of more than 150mg need to be given subcutaneously at different sites in two or more times

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ age ≤50 years, and in good health;
* 40kg ≤ weight ≤100kg , and body mass index is within the range of 18 - 28 kg/m^2 (including 18 kg/m^2 and 28 kg/m^2);
* No parental scheme from the screening period to 6 months after the study period.

Exclusion Criteria:

* Participants have abnormal physical and auxiliary examination results with clinical significance;
* History of cardiovascular, liver, kidney, digestive, blood, nervous system and allergic diseases, mental and metabolic disorders, acute or chronic bronchospastic disease;
* Smoking more than 5 cigarettes per day;
* Participants who use any prescription drugs within 4 weeks prior dosing, or over-the-counter medication within 2 weeks prior to dosing. Participants who receive treatment of any biologics within three months prior to dosing. Participants who receive (attenuated) live vaccines within six months prior to dosing;
* Participation in any clinical investigation within 3 months prior to dosing;
* Donation or loss of 400 mL or more of blood within 3 months prior to dosing; donation or loss of 200 mL or more of blood within 4 weeks prior to dosing; or donation of component blood within 2 weeks prior to dosing;
* Tuberculosis symptoms, contact with patients with suspected tuberculosis symptoms
* Positive results in Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, Syphilis antibody or HIV antibody;
* Clinically significant acute infection within 2 weeks prior to dosing;
* Current or previous drug or alcohol abuse;
* Other conditions in which the investigator preclude enrollment into the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Maximum observed serum Genakumab concentration | Baseline, 0.5h, 1h, 2h, 4h, 8h, 12h, 24h, 48h, 72h, 96h, 168h, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71, Day 85, Day 99, Day 113 after administration
Area under the serum Genakumab concentration-time curve | Baseline, 0.5h, 1h, 2h, 4h, 8h, 12h, 24h, 48h, 72h, 96h, 168h, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71, Day 85, Day 99, Day 113 after administration
Measurement of the serum IL-1β for pharmacodynamics study | Baseline, 0.5h, 1h, 2h, 4h, 8h, 12h, 24h, 48h, 72h, 96h, 168h, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71, Day 85, Day 99, Day 113 after administration

SECONDARY OUTCOMES:
The frequency of adverse events (AE) | From screening to follow-up period (up to day 22)

CONTACTS AND LOCATIONS:
Overall Officials: Rui Chen, Principal Investigator — Clinical Pharmacology Research Center of Peking Union Medical College Hospital
Locations (1):
- Clinical Pharmacology Research Center of Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Liu H, Yuan Y, Tian W, Luo T, Xu Q, Zhu X, Chen R. Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Firsekibart, an Anti-interleukin-1beta Monoclonal Antibody, in Healthy Chinese Participants: A Randomized, Double-Blind, Placebo-Controlled Phase 1 Study. Adv Ther. 2025 Sep;42(9):4611-4625. doi: 10.1007/s12325-025-03279-4. Epub 2025 Jul 25. PMID 40711661